CLINICAL TRIAL: NCT04097691
Title: Injection of Subcutaneous Glucose 10% in Small Shots is Effective in the Treatment of Diabetic Neuropathic Pain
Status: Completed | Type: Observational
Sponsor: Ministry of Health and Population, Egypt (Other Government)
Responsible Party: Principal Investigator, mahmoud younis, Principal Investigator, Ministry of Health and Population, Egypt
Other Study IDs: mahmoudyounis
Record Dates: First submitted 2019-09-13; First posted 2019-09-20 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Painful Diabetic Neuropathy
Keywords: diabetes mellitus; diabetic neuropathy; pain; glucose 10%
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- on subcutaneous glucose: this group was on subcutaneous glucose 0.5 ml per site around subcutaneous nerves in the foot region both on palm and sole.which is repeated every 2 weeks for 2 months.
  Interventions: Drug: GLUCOSE 10%
- control(not receiving treatment): the second group is considered as control.received no treatment.
  Interventions: Drug: GLUCOSE 10%

INTERVENTIONS:
Drug: GLUCOSE 10% — subcutaneous glucose 0.5 ml per site around subcutaneous nerves
  Other Names: dextrose 10%

SUMMARY:
Observational cohort prospective study with the following of 100 patients of type 1 and type 2 diabetes mellitus in 2 groups each group 50 patients, each group 30 males, and 20 females,35 patients with type 2 diabetes and 15 patients type 1 diabetes all have diabetic peripheral neuropathy, the second group is considered as control.

DETAILED DESCRIPTION:
Observational cohort prospective study with the following of 100 patients of type 1 and type 2 diabetes mellitus in 2 groups each group 50 patients, each group 30 males, and 20 females,35 patients with type 2 diabetes and 15 patients type 1 diabetes all have diabetic peripheral neuropathy, the second group is considered as control. the ages of all patients are between 20 and 50 years.

The first group was on subcutaneous glucose 0.5 ml per site around subcutaneous nerves in the foot region both on palm and sole.which is repeated every 2 weeks for 2 months.

Pain severity was evaluated by using the Visual Analogue Scale (VAS) which is a numerical rating scales, with a straight horizontal line of 100 mm. which is directed from the left with severe pain to the right with no pain. 1-3 = mild pain,4-6 = moderate pain,7-10 = severe pain.

The evaluation of neuropathy was done by using the Michigan Neuropathy Screening Instrument (MNSI) after translation to the Arabic language.which consists a 15 self-administered questionnaires and examination lower extremities which comprise inspection and examination of vibratory senses and ankle reflexes. A score which is more than 7 was suggested to be abnormal.

ELIGIBILITY:
Inclusion Criteria:

1. patients 20 years to 50 years with type 1 or type 2 diabetes who have symptoms of symmetrical peripheral neuropathic pain.
2. female Patients are not pregnant.
3. Patient has a pain score of at least 5 on the Visual Analogue Scale (VAS).
4. Patients are on their antidiabetes medication.
5. patents are not on any medication for peripheral neuropathy.
6. Patient must be able to complete questions on the Michigan Neuropathy Screening Instrument (MNSI).

Exclusion Criteria:

1. Patient has conditions that could affect the evaluation of painful DPN, or non-diabetic neurologic disorders.
2. Patient has skin conditions in the area affected by the neuropathy that could alter sensation.
3. Patient with history of drug abuse.
4. patients on any drug for diabetic neuropathy like pregabalin or gabapentin. No side effects were monitored during the period of treatment.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 100 patients of type 1 and type 2 diabetes mellitus in 2 groups each group 50 patients, each group 30 males, and 20 females,35 patients with type 2 diabetes and 15 patients type 1 diabetes all have diabetic peripheral neuropathy, the second group is considered as control. the ages of all patients are between 20 and 50 years.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-07-14 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

PRIMARY OUTCOMES:
Injection of subcutaneous glucose 10% in small shots is effective in treatment of diabetic neuropathic pain measured the Visual Analogue Scale (VAS) | from baseline to 2 months
  Pain severity was evaluated by using the Visual Analogue Scale (VAS) which is a numerical rating scale, with a straight horizontal line of 100 mm. which is directed from the left with severe pain to the right with no pain. 1-3 = mild pain,4-6 = moderate pain,7-10 = severe pain.
Injection of subcutaneous glucose 10% in small shots is effective in improving neuropathic signs using the Michigan Neuropathy Screening Instrument (MNSI) | from baseline to 2 months
  The evaluation of neuropathy was done by using the Michigan Neuropathy Screening Instrument (MNSI) after translation to the Arabic language. Which consists a 15 self-administered questionnaires and examination of lower extremities which comprise inspection and examination of vibratory senses and ankle reflexes. A score which is more than 7 was suggested to be abnormal.

CONTACTS AND LOCATIONS:
Locations (1):
- Mahmoud Younis, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No